CLINICAL TRIAL: NCT01350908
Title: Development and Validation of a Circulating Tumor DNA Detection Technique in Patients With Ovarian Cancer
Brief Title: Study of Circulating Tumoral DNA in Ovarian Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IC2010-03
Record Dates: First submitted 2011-05-06; First posted 2011-05-10 (Estimated); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Blood sampling (Other)
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — 30mL of peripherical blood will be collected specially for the study. It's an additional blood sampling compare to the normal follow up of the patient.

SUMMARY:
Circulating tumor DNA detection and quantification in patients with ovarian cancer.

DETAILED DESCRIPTION:
Technique development:

In a first step, the different available techniques will be evaluated for specificity and sensibility using serial dilutions of cell lines with or without TP53 mutation.

Validation:

The tumor DNA detection rate will be estimated from patient's blood with ovarian cancer.

The investigators will study 25 patients to obtain at least 15 patients bearing a TP53 mutation that could be characterized in the primitive tumor or metastasis. With those 15 patients, the investigators will determine the most sensitive technique and the best cost/efficiency ratio.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18 years.
* Patient with invasive ovarian cancer stage II to IV from FIGO classification.
* Patient treated by surgery.
* Patient with tumor or metastasis available for TP53 status characterization
* Patient able to stand a blood collection.
* Signed written informed consent approved by AFSSAPS and CPP.

Exclusion Criteria:

* Patient without social protection / insurance.
* Borderline ovarian tumor.
* Non carcinoma ovarian tumor
* Patient with invasive ovarian cancer 5 years before diagnosis
* Current pregnancy and lactation.
* All social, medical, psychological, situations making the study impossible.
* Person deprived of liberty.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-04; Primary Completion 2015-01 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Assessment and development of circulating tumor DNA detection techniques | 2 years
  Quantification of circulating tumor DNA in blood samples. Results expressed in number of samples where circulating DNA is present.

SECONDARY OUTCOMES:
Comparison of the detection techniques (PAP (pyrophosphorolysis activated polymerisation), BEAMing, NGS(Next sequencing generation) with regards to feasibility, robustness, sensitivity and cost. | 2 years
  The methods of detection which will be used such as the BEAMing, the PAP(pyrophosphorolysis activated polymerization) and the NGS(next sequencing generation is techniques of a big specificity capable of detecting a mutant copy among 1.104 wild copies for the BEAMing, 2.109 for the PAP and 1.105 for the NGS. The sensibility of these techniques is limited by the quantity of genomic DNA which we can extract from the sample of blood.

CONTACTS AND LOCATIONS:
Overall Officials: LANTZ Olivier, MD, Principal Investigator — Institut Curie
Locations (1):
- Institut Curie, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).